CLINICAL TRIAL: NCT00950716
Title: Peer Support, Empowerment and Remote Communication Linked by Information Technology (PEARL): A Multi-Component Program to Improve Community-Based Diabetes Care
Brief Title: PEARL Program: Empowerment Program for Patients With Type 2 Diabetes (HK4)
Acronym: PEARL
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: Asia Diabetes Foundation (Other)
Responsible Party: Principal Investigator, Juliana Chan, Chair Professor of Medicine and Therapeutics, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: CRE-2009-079
Record Dates: First submitted 2009-07-31; First posted 2009-08-03 (Estimated); Last update posted 2015-08-25 (Estimated); Status verified 2015-08

CONDITIONS: Diabetes
Keywords: type II diabetes; peer support; empowerment
MeSH Terms: conditions — Diabetes Mellitus; Diabetes Mellitus, Type 2; Empowerment

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Usual care (Active Comparator): The 'control arm' will receive standard usual care with clinicians' follow-up and referral with education to diabetes nurses if deemed necessary at in-charge clinicians' discretion.
  Interventions: Behavioral: Usual Care
- Patient Peer Support and Empowerment (Active Comparator): 30 mentors are themselves diabetes patients who have good self care and are motivated to support their peers. The mentors will be trained to deliver peer support intervention under supervision by a program manager. The 300 diabetes patients (mentees) randomized to the peer support group are the intervention targets of these 30 mentors. Telephone-Linked-Communication (TLC) system will be a tool of the mentors for education to the mentees. TLC system utilizes an automatic, interactive, computer-controlled telephone system to monitor and promote diabetes self-management.
  Interventions: Behavioral: Patient Peer Support and Empowerment

INTERVENTIONS:
Behavioral: Patient Peer Support and Empowerment — 30 mentors are themselves diabetes patients who have good self care and are motivated to support their peers. The mentors will be trained to deliver peer support intervention under supervision by a program manager. The 300 diabetes patients (mentees) randomized to the peer support group are the intervention targets of these 30 mentors. Telephone-Linked-Communication (TLC) system will be a tool of the mentors for education to the mentees. TLC system utilizes an automatic, interactive, computer-controlled telephone system to monitor and promote diabetes self-management.
  Arms: Patient Peer Support and Empowerment
Behavioral: Usual Care — Subjects in Usual CAre will receive standard care with clinicians' usual follow-up and referral with education to diabetes nurses if deemed necessary at in-charge clinicians' discretion.
  Arms: Usual care

SUMMARY:
Quality diabetes care requires informed-decisions of motivated care providers and diabetes patients. The investigators aim to use peer support and information technology to facilitate care providers to implement structured care and empower diabetes patients acquire self-management skills in a multi-component program.

The investigators will make use of the following tools: (1) The Joint Asia Diabetes Evaluation (JADE) Program. JADE Program uses a web-based electronic portal to establish a registry and stratify diabetes patients to care protocols based on their risk profiles with features of decision support and data management. (2) The Australasian Telephone Linked Care (TLC) system. TLC system utilizes an automatic, interactive, computer-controlled telephone system to monitor and promote diabetes self-management.

Amongst 600 diabetes patients receiving structured care in Hong Kong through the JADE Program, half of them will be randomized to receive peer support (n=300) including personal coaching by 30 trained mentors (1 mentor to 10 diabetes patients or mentees) through regular phone calls and sharing sessions, and the other half (n=300) will continue the usual diabetes care in their clinic. The 30 mentors are themselves diabetes patients who have good self care and are motivated to support their peers. The mentors will be trained to deliver peer support intervention under supervision by a program manager. The 300 diabetes patients (mentees) randomized to the peer support group are the intervention targets of these 30 mentors. They will be reminded to use the TLC for knowledge enhancement and motivational support.

The investigators will analyse the changes in risk factor control (blood glucose parameters, blood pressure, body weight, lipids), quality of life and cognitive-psychological-behavioral parameters after 12 months. Effects of various components of peer support on these outcomes as well as user acceptability and cost-effectiveness of these programs will be examined.

The investigators will test the hypothesis that in a multi-component program, the use of a peer support program delivered by diabetes patient-mentors, to influence and motivate other diabetes patients receiving structured care made possible through a web-based disease management program, delivered by a doctor-nurse team, will further improve metabolic control, QOL and self care compared to diabetes patients receiving the same standard of care.

DETAILED DESCRIPTION:
In this global epidemic of diabetes and obesity, more than 60% of affected people will come from Asia with the most rapid increase in the young to middle aged group. This rapid increase in young onset diabetes will have major implications on health care costs, quality of life and societal productivity. Despite the amassing body of evidence supporting the highly preventable nature of diabetes and associated complications, there are multiple barriers in the implementation of quality diabetes care. Apart from issues relating to health care systems and reimbursement, the silent nature of diabetes and associated complications as well as the complex nature of care protocols which requires frequent evaluation of clinical and laboratory parameters and the need for diabetes patients to adhere to long term medications and self care are important factors.

Diabetes is a prototype of chronic diseases covering the full spectrum of health promotion, disease prevention, management and rehabilitation. To achieve these inter-dependent goals, multiple levels of expertise and support are needed to preserve health, prevent complications and enhance quality of life. A successful diabetes care program depends on informed decisions of motivated care providers and diabetes patients who require periodic comprehensive assessments for risk stratification and individualized management which include education, assessments, feedback and technologies.

According to the International Diabetes Federation (IDF) global guidelines (www.idf.org), standard diabetes care include the delivery of culturally sensitive care, cultivation of relationship between care providers and diabetes patients, offer of annual surveillance, goal setting on care plans and targets, adherence to protocol, provision of access to patient-centred care using a multidisciplinary team, establishment of a registry for recall, provision of telephone contact and patient support group and a quality assurance and improvement program. Comprehensive care includes all components of standard of care together with access of diabetes patients to their own data and decision support.

To achieve this ambitious goal, delivery of chronic care must be integrated with effective self management on a long term basis. People with diabetes need to acquire knowledge, skills and attitudes to exercise self discipline on food choices, physical activity, self monitoring and management of negative emotions. To this end, experts have identified 6 key resources and support for self management including 1) individualized assessment, 2) collaborative goal setting, 3) skills enhancement, 4) follow-up and support, 5) access to resources, and 6) continuity of quality clinical care.

However, most studies which use cognitive and psychological strategies to effect behavioral changes have reported high rates of relapse despite initial success, often due to negative external or social influences. Thus, to enhance self management, there is a need to take into consideration both internal needs (assessment of individual needs, learning skills and goal setting) and external support (e.g. families, organizations, neighborhoods, and communities) to encourage and reinforce the use of learned skills to sustain positive behavior and self management on a long term basis. Adding to these emerging concepts in behavioral medicine is equifinality, i.e. diverse approaches may achieve similar end. Thus, a multi-component program offering a broad range of intervention approaches may tailor the pluralistic needs of people with diabetes or chronic disease.

Aims of the Study:

1. To quantify the impacts of peer support on self management skills, quality of life (QOL) and cognitive-psychological-behavioral parameter.
2. To quantify effects of various components of self management skills and cognitive- psychological-behavioral parameters on metabolic control, care processes and QOL.
3. To examine the user acceptability (including health care team and diabetes patients) and cost effectiveness of this multi-component system in improving diabetes care in the community..

ELIGIBILITY:
Inclusion Criteria:

* 1) Type 2 diabetic patients with medium or moderate risk for complications (stratified by JADE Program, Care Levels 2 to 4) and followed up 3-4 monthly according to the JADE Program. Based on our 6000-patient registry, these risk levels clearly separate diabetes patients based on risk of future clinical events.
* 2) Men/women aged 18-70 years (inclusive), functionally independent and with informed written consent.

Exclusion Criteria:

* 1) Patients with one or no risk factors (low risk, Care Level 1 by JADE Program) as stratified by the JADE Risk Engine.

  2) Patients with reduced life expectancy and unstable mood or major psychiatric conditions.

  3) Patients who cannot communicate in Chinese language.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 632 (Actual)
Dates: Start 2009-09; Primary Completion 2015-02 (Actual); Study Completion 2015-02 (Actual)

PRIMARY OUTCOMES:
Glycemic control | one year
Body weight | one year
Blood pressure | one year
Lipid levels | one year

SECONDARY OUTCOMES:
Cognitive-psychological-behavioral assessments: a) Depression Anxiety and Stress Scale (DASS21). b) Diabetes Empowerment Scale (C-DES). c) Summary of Diabetes Self Care Activities (SDSCA, Chinese version). | One year

CONTACTS AND LOCATIONS:
Locations (1):
- Asia Diabetes Foundation, Hong Kong, China

REFERENCES:
- [Derived] Yeung RO, Cai JH, Zhang Y, Luk AO, Pan JH, Yin J, Ozaki R, Kong APS, Ma R, So WY, Tsang CC, Lau KP, Fisher E, Goggins W, Oldenburg B, Chan J. Determinants of hospitalization in Chinese patients with type 2 diabetes receiving a peer support intervention and JADE integrated care: the PEARL randomised controlled trial. Clin Diabetes Endocrinol. 2018 Mar 7;4:5. doi: 10.1186/s40842-018-0055-6. eCollection 2018. PMID 29541481
- [Derived] Chan JC, Sui Y, Oldenburg B, Zhang Y, Chung HH, Goggins W, Au S, Brown N, Ozaki R, Wong RY, Ko GT, Fisher E; JADE and PEARL Project Team. Effects of telephone-based peer support in patients with type 2 diabetes mellitus receiving integrated care: a randomized clinical trial. JAMA Intern Med. 2014 Jun;174(6):972-81. doi: 10.1001/jamainternmed.2014.655. PMID 24781960
- See also: details of the Peers for Progress Grant and its aims; and the grantees in 2009 — http://www.peersforprogress.org/
- See also: Works, including PEARL program, of Asia Diabetes Foundation — http://www.adf.org.hk